CLINICAL TRIAL: NCT00425022
Title: Feasibility of VATS(Video-Assisted Thoracoscopic Surgery) Lobectomy for Clinical Stage IB or II Non-Small Cell Lung Cancer
Brief Title: VATS Lobectomy for Clinical Stage IB or II Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-223
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Thoracic Surgery, Video-Assisted
Keywords: lung cancer; video-assisted thoracic surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Thoracoscopy

INTERVENTIONS:
Procedure: thoracoscopy

SUMMARY:
To examine the feasibility of VATS lobectomy for clinical stage IB or II non-small cell lung cancer. Success is defined as VATS lobectomy without conversion. If success rate over 90%, VATS lobectomy is considered as feasible procedures for clinical stage IB or II non-small cell lung cancer

DETAILED DESCRIPTION:
Video-assisted or minimally invasive surgery has become the standard approach for many abdominal surgical operations such as cholecystectomy and fundoplication. With respect to the thorax, video-assisted thoracoscopic surgery(VATS) is the accepted technique for biopsy of the lung and pleura and surgical treatment of pneumothorax.Thoracoscopic, also termed video-assisted thoracoscopic lobectomy has become accepted as a safe and effective procedure to treat early-stage non-small cell lung cancer (NSCLC). Several pilot series of thoracoscopic lobectomy in stage I lung cancer patients have been reported, demonstrating low complication rates and effective short-term and long-term oncologic results. With increasing experience, the indications for thoracoscopic lobectomy have been expanded. Single and Multi-institutional studies have demonstrated that thoracoscopic lobectomy is not only a safe and feasible technique, but is also associated with decreased morbidity, including shorter length of hospitalization and chest tube duration, decreased postoperative pain, improved preservation of pulmonary function, reduced inflammatory response as measured by lower postoperative cytokine levels, and shorter recovery time, as compared with conventional thoracotomy. The advantages of thoracoscopic lobectomy have been demonstrated in patients with clinical stage I NSCLC, and this strategy has been found to be particularly useful for specific subsets of patients such as the elderly and those patients with poor performance status.

The purpose of this study is to know whether VATS lobectomy for clinical stage IB or II non-small cell lung cancer is possible.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of non-small cell lung cancer.
2. Clinical stage IB or II, according to the American Joint Committee on Cancer (AJCC).
3. Tumor ≤ 6 cm in size amenable to surgical resection.
4. Including clinical IB or II NSCLC after neoadjuvant therapy
5. Performance status of 0-1 on ECOG scale.
6. At least 18 years old.
7. Patient compliance that allows adequate follow-up.
8. Medical fitness of patients adequate for radical NSCLC surgery.
9. Adequate organ function including the following:Adequate hematologic function: WBC count ³ 4,000/uL, absolute neutrophil count (ANC) ³ 1,500/uL, platelet count ³ 100,000/uL, and hemoglobin ³ 10 gm/dL.Adequate hepatic function: bilirubin £ 1.5 x UNL, ALT or AST £ 2.5 x UNL.Adequate renal function: creatinine £ 1.5mg/dL.
10. Signed informed consent from patient or legal representative.
11. Patients with reproductive potential must use an approved contraceptive method during and for 3 months after the study. Females with childbearing potential must have a negative urine hCG test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Metastatic disease in workup
2. Any T3, T4 lesion or N2, N3 lesion
3. Concurrent administration of other tumor therapy, including radiotherapy, immunotherapy except chemotherapy.
4. Active uncontrolled infection.
5. Serious concomitant disorders that would compromise the safety of patient or compromise the patient's ability to tolerate therapy.
6. Significant neurological or mental disorder.
7. Previous history of malignancy in any organ
8. Pregnant or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-01

PRIMARY OUTCOMES:
To examine the feasibility of VATS lobectomy for clinical stage IB or II non-small cell lung cancer.
Success is defined as VATS lobectomy without conversion.
If success rate over 90%, VATS lobectomy is considered as feasible procedures for clinical stage IB or II non-small cell lung cancer

SECONDARY OUTCOMES:
To evaluate the number of dissected lymph nodes and the rate of contamination during lymph node dissection according to the lymph node stations under VATS
To estimate the reccurrence rate (locoregional and distant metastasis)
To estimate the overall survival
To evaluate the intraoperative(surgical duration, estimated blood loss) and postoperative variables(mortality, morbidity, chest tube drainage duration, wound pain, hospital stay)
To evaluate inflammatory mediators after VATS

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Sung Lee, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- See also: Video presentation about complete lymph node dissection under VATS — http://www.ctsnet.org